CLINICAL TRIAL: NCT04288492
Title: The Effect of Respiratory Exercise Using Preoperative Biofeedback on Postoperative Pain
Brief Title: Effect of Biofeedback on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Gyeongsang National University Hospital (Other)
Responsible Party: Principal Investigator, BON WOOK KOO, assistnat professosr, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: biofeedback112233
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Pain
Keywords: Respiratory biofeedback; Postpoerative Pain; Preoperative Anxiety
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biofeedback (Experimental): Respiratory exercise using biofeedback device(ResCalm) 2-3 times / day for 3 minutes until discharge from hospital, once in recovery room before surgery
  Interventions: Behavioral: Respiratory biofeedback
- general (No Intervention): General surgical schedule without control exercise

INTERVENTIONS:
Behavioral: Respiratory biofeedback — Repeat the inspiration and exhalation breaths for a fixed period of time using a biofeedback device (ResCalm)
  Arms: biofeedback

SUMMARY:
This study is a multi-center, randomized, controlled, double-blinded, and parallel design study. A total of 106 patients were decided to be recruited considering a 10% dropout rate. Patients are randomizes to perform or not respiratory exercises using biofeedback device(ResCalm). The randomization numbers are generated using a computer-generated randomization code and are sealed in the opaque envelope until they are handed over to anesthesiologist in charge of patient management. Record patient preoperative t anxiety, postoperative pain, and pain medication use. Patient aged 19-64 yr, ASA class 1 or 2, and are scheduled for elective laparoscopic cholecystectomy are included. Patients who were unable to perform self breathing at regular intervals were excluded.

DETAILED DESCRIPTION:
1. Assignment of experimental groups

   Group A: Respiratory exercise using respiratory biofeedback device(ResCalm) is applied 2-3 times / day for 3 minutes until discharge from hospital and once in the recovery room before surgery.

   Group B: General surgery schedule without control exercise.

   All patients measure STAI(state trait anxiety inventory) at the operating room entrance on the day of surgery.
2. anesthesia methods Intravenous anesthesia is performed using the target injection concentration control method. As an anesthetic, propofol / remifentanil / rocuronium is used. The artificial ventilation method is a pressure-controlled ventilation method, which maintains an appropriate pressure and performs anesthesia.
3. postoperative care After anesthesia, the patient wakes up and transfers to the recovery room to encourage self-breathing exercise. After entering the recovery room, the patient's vital signs (average blood pressure, heart rate, oxygen saturation) and analgesic use are checked immediately before leaving.

The investigators check for the presence of pulmonary complications, visual analog scale (VAS), analgesic use, and hospital patient satisfaction for 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 19 and 64 years of age with ASA class I, II who underwent regular laparoscopic cholecystectomy under general anesthesia.

Exclusion Criteria:

* Seniors 65 years of age or older or minors under 19 years of age
* ASA (American Society of Anesthesiologists) class ≥ III
* Difficulties in proper cooperation with diseases such as Alzheimer dementia, cognitive disorders, and psychopathy
* Patients with respiratory diseases such as Asthma, Pnuemonia
* Patients with incomplete airway due to pulmonary resection, airway surgery, mouth or nose surgery

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Total score of STAI(state-trait anxiety inventory) | 20 minutes before the anesthesia started.
  Preoperative anxiety state is measured using STAI(state-trait anxiety inventory): Total score of 40 questions.
  Each question is consisted as follows
  1: not at all 2: a little 3: somewhat 4: very much so minimal: 40 maximum: 160

SECONDARY OUTCOMES:
Total amount of cumulative analgesics | 24 hours after the anesthesia finished.
  total amount of analgesics are measured for 24 hours after surgery.
The rate of Pulmonary complication | 24 hours after the anesthesia finished.
  medical record is checked after operation
The score of pain | 24 hours after the anesthesia finished.
  VAS(visual analog scale) measurement for 24 hours after surgery(0-10) 0: no pain 10: severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Bon Wook Koo, MD, Study Director — SNUBH
Locations (1):
- Bon Wook Koo, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No